CLINICAL TRIAL: NCT04916132
Title: Biopsy-proven Diabetic Nephropathy in People With Type 2 Diabetes. Prevalence and Predictive Factors
Brief Title: Diabetic Nephropathy in People With Diabetes. Prevalence and Predictive Factors
Acronym: PRIMETIME2
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hillerod Hospital, Denmark (Other); Zealand University Hospital (Other); Holbaek Sygehus (Other); Slagelse Sygehus (Other); Nykøbing Falster County Hospital (Other); Aarhus University Hospital (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other); Novo Nordisk A/S (Industry); Gubra ApS (Unknown); Odense University Hospital (Other); Aalborg University Hospital (Other); Gødstrup Hospital (Other); Steno Diabetes Center Copenhagen (Other); Steno Diabetes Center Sjaelland (Other Government); Steno Diabetes Center Nordjylland (Other); Michigan Kidney Translational Medical Center (Unknown)
Responsible Party: Principal Investigator, Marie Møller, MD, PhD-student, Herlev Hospital
Other Study IDs: PRIMETIME2; H-20080050 (Other: National Ethical Committee)
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Albuminuria; Diabetic Kidney Disease; Diabetic Nephropathies; Diabetes type2; Molecular Sequence Variation; Kidney Biopsy
Keywords: diabetic nephropaty; precision medicine; kidney biopsy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Kidney Biopsy (histological and RNA-sequencing) Blood (proteomics, metabolomics and wholegenome sequencing) Urine (Proteomics and metabolomics) Faecal and salvia samples (analysis om the microbiom)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peolpe with T2DM and albuminuria: Prospectively we will collect research kidney biopsies and other biomarkers from blood, faeces, urine, proteomic- and metabolomic profiles and DNA-variants. The biopsies will be thoroughly investigated with cutting-edge molecular technologies and associated to the biomarkers, disease course and clinical outcome.
  Interventions: Procedure: Kidney Biopsy

INTERVENTIONS:
Procedure: Kidney Biopsy — Harvesting of kidney tissue from people with type 2 diabetes and albuminuria for subsequent analysis

SUMMARY:
a prospective, observational, multi-center study with a cohort of 300 patients with Type 2 diabetes and macroalbuminuria. Prospectively we will collect kidney biopsies and analyse the transciptome of the kidney tissue and other biomarkers from blood, faeces, urine, proteomic- and metabolomic profiles and DNA-variants. Thereby we hope to be able to discover molecular and clinical profiles, that can help us in the diagnosis of DKD, and to identify different risks of progression that can benefit from different forms of personalized treatment.

DETAILED DESCRIPTION:
The PRIMETIME project is made to bring together molecular, translational and clinical scientists to create collaborations and build a scientific bridge between diabetology, nephrology, clinical biochemistry, and pathology. The ultimately goal is to bring forward an improved understanding of the most frequent cause of end stage renal disease: DKD. We aim to improve the diagnostic accuracy as well as the treatment precision by investigating in detail the features of histology and protein expression in both retrospective(WP1) and prospective(WP2) kidney biopsy material.

PRIMETIME WP2 is a prospective, observational, multi-center study with a cohort of 300 patients. We plan to create a systematically unselected cohort of patients with Type2 diabetes and macroalbuminuria as a sign of kidney injury. Prospectively we will collect research kidney biopsies and other biomarkers from blood, faeces, urine, proteomic- and metabolomic profiles and DNA-variants. The biopsies will be thoroughly investigated with cutting-edge molecular technologies and associated to the biomarkers, disease course and clinical outcome. The participants will afterward be followed in 20 years.Thereby we hope to be able to discover molecular and clinical profiles, that can help us in the diagnosis of DKD, and to identify different risks of progression that can benefit from different forms of personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* Diagnosis with T2DM according to the American diabetes Association (20)
* eGFR >30 mL/min/1.73 m2 (maximum six months old)
* urine-albumin/creatinine-ratio (uACR) > 700 mg/g or 24 hours urine albumin >700 mg on more than one measurement

Exclusion Criteria:

* Signs of acute kidney failure according to the KDIGO classification (21) at the time for kidney biopsy or the last 6 months before kidney biopsy
* Factors that increases the risk of complications due to kidney biopsy:

  * Hemoglobin < 6 mmol/L
  * INR >1,4 at the time for biopsy
  * Platelet count < 100 x 109/l
  * Uncontrolled high blood pressure (defined as systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg)
  * Only one functioning kidney
  * Evidence of urinary tract obstruction or hydronephrosis at the time of biopsy
  * Multiple bilateral kidney cysts
  * Kidney infection, peri-renal infection, or cutaneous infection that overlies the kidney at time for biopsy
  * Unwilling to receive blood transfusion
  * Unable to lie flat in bed six hours after biopsy
  * Any other contra-indications for percutaneous kidney biopsy according to local clinical guidelines
* Unable to understand written and oral information
* Kidney transplant recipient
* Previous medical kidney biopsy
* Women who are pregnant or planning to become pregnant before the kidney biopsy is performed
* Treatment with Marcoumar (all other anticoagulants are accepted)
* High thromboembolic risk combined with held in anticoagulation therapy according to the report "Perioperative regulation of antithrombotic treatment" (PRAB) (22)

  * mechanical heart valve
  * atrial fibrillation AND CHA2DS2-VASc> 5 and/or stroke within the last three months
  * recurrent venous thromboembolism OR venous thromboembolism within the last three months
  * less than 6 weeks after uncomplicated Acute Coronary Syndrome (ACS) with or without revascularization (Percutaneous Coronary Intervention (PCI)) with Bare Metal Stents (BMS) or Coronary Artery Bypass Grafting (CABG))
  * less than 3 months after uncomplicated ACS with revascularization (PCI with Drug Eluting Stent (DES))
  * less than 9-12 months after complicated ACS (e.g. reinfarction or stent thrombosis)
  * less than 1 month after revascularization in individuals with stable Coronary Artery Disease (CAD) (PCI with BMS or CABG)
  * less than 3 months after revascularization in individuals with stable CAD (PCI with DES)
  * less than 3 months after stroke, or Transient Ischemic Attack (TIA)
* Inability to withdraw nonsteroidal anti-inflammatory drugs (NSAID) 7 days before biopsy

If a participant meets one or more exclusion criteria, that are reversible, the participant can be rescreened later on, to evaluate whether or not the participant now is qualified for participation.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with type 2 diabetes, albuminuria and eGFR > 30 who are willing to undergo a kidney biopsy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence | From baseline to end inclusion (3 years)
  To investigate the prevalence of biopsy-proven diabetic nephropathy in individuals with T2DM with severe albuminuria; urine albumin/creatinine ratio (UACR) >700 mg/g.

SECONDARY OUTCOMES:
Improved clinical diagnosis | From baseline to end inclusion (3 years)
  To investigate whether clinical variables, transcriptomic, proteomic and/or metabolomic profiles as well as genetic variation can predict the presence of diabetic nephropathy in a kidney biopsy.
diabetic retinopathy | From baseline to end inclusion (3 years)
  To describe the sensitivity and specificity of diabetic retinopathy in predicting biopsy-proven diabetic nephropathy
Kidney Biopsy | From baseline to end of followup (20 years)
  describe the prognostic value of different histological and molecular findings on kidney biopsy in individuals with biopsy-proven diabetic nephropathy
non-diabetic nephropathy vs. biopsy-proven diabetic nephropathy | From baseline to end of followup (20 years)
  describe the prognostic value of different histological and molecular findings on the kidney biopsy in individuals with non-diabetic nephropathy compared to biopsy-proven diabetic nephropathy.
proteomic and metabolomic | From baseline to end of followup (20 years)
  describe the prognostic value of the proteomic and metabolomic profiles in biopsy-proven diabetic nephropathy.
genetic variants | From baseline to end of followup (20 years)
  describe the prognostic value of different forms of genetic variation in biopsy-proven diabetic nephropathy
Microbiome | From baseline to end of followup (20 years)
  describe the prognostic value of different compositions of the microbiome and its relation to biopsy and clinical findings
Annual changes in kidney status | From baseline to end of followup (20 years)
  Annual changes in kidney status (defined by yes/no: initiation of dialysis, kidney transplantation, renal death or decrease in eGFR > 40 % compared to eGFR at baseline)
Annual decline in eGRF | From baseline to end of followup (20 years)
  Annual decline in eGRF
Annual changes in albuminuria. | From baseline to end of followup (20 years)
  Annual changes in albuminuria.
Annual events of cardiovascular disease | From baseline to end of followup (20 years)
  Events of cardiovascular disease (fatal CV events, non-fatal stroke, non-fatal myocardial infarction, hospitalization for heart failure, PCI or bypass surgery (heart or legs), amputations due to ischemia, and unstable angina)
Death | From baseline to end of followup (20 years)
  Death (any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Persson, MD, PhD, Study Chair — Steno Diabetes Center Copenhagen
Locations (13):
- Denmark (13):
  - Aarhus Universitetshospital, Skejby, Skejby, Aarhus
  - Steno Diabetes Center Copenhagen, Copenhagen, Gentofte
  - Kristine D Schandorff, Hillerød, Hillerød
  - Holbæk Hospital, Holbæk, Holbæk
  - Rigshospitalet, Copenhagen, København Ø
  - Sjællands Universitetshospital, Køge, Køge, Køge
  - Nykøbing Falster Sygehus, Nykøbing Falster, Nykøbing F
  - Sjællands Universitetshospital, Roskilde, Roskilde, Roskilde
  - Slagelse Sygehus, Slagelse, Slagelse
  - Aalborg universitetshospital, Aalborg
  - Regionshospitalet Gødstrup, Gødstrup
  - Herlev Hospital, Herlev
  - Odense universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided
This topic is still up for discussion. We do plan to share most of the data, but how, time and place are still undecided

REFERENCES:
- [Derived] Moller M, Borg R, Bressendorff I, Fink LN, Gravesen E, Jensen KH, Hansen T, Krustrup D, Persson F, Rossing P, Sembach FE, Thuesen ACB, Hansen D. Rationale and design of a prospective, clinical study of kidney biopsies in people with type 2 diabetes and severely increased albuminuria (the PRIMETIME 2 study). BMJ Open. 2023 Jun 6;13(6):e072216. doi: 10.1136/bmjopen-2023-072216. PMID 37280026